CLINICAL TRIAL: NCT01334372
Title: Intensive Outpatient Treatment for Suicidal Veterans: A Randomized Clinical Trial and Feasibility Investigation
Brief Title: Intensive Outpatient Treatment for Suicidal Veterans
Acronym: CAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); The Catholic University of America (Other)
Responsible Party: Lisa Brenner, VISN 19 Mental Illness Research, Education, and Clinical Center
Other Study IDs: 06-1058
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Suicidality
Keywords: suicide; veterans; assessment; CAMS
MeSH Terms: conditions — Suicidal Ideation; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (No Intervention): Treatment as usual (TAU) outpatient care will consist of existing outpatient clinical practices utilized in the Mental Health Clinic.
- CAMS (Experimental): First, as discussed above, suicidality is the focus of treatment rather than one of many symptoms being treated. Second is the emphasis on patient and therapist collaborating on treatment rather than the therapist dictating how therapy progresses. Beyond those two basic tenets, each therapist is free to utilize their current clinical skills to conduct psychotherapy.
  Interventions: Behavioral: CAMS

INTERVENTIONS:
Behavioral: CAMS — First, as discussed above, suicidality is the focus of treatment rather than one of many symptoms being treated. Second is the emphasis on patient and therapist collaborating on treatment rather than the therapist dictating how therapy progresses. Beyond those two basic tenets, each therapist is free to utilize their current clinical skills to conduct psychotherapy.
  Arms: CAMS

SUMMARY:
This investigation is a feasibility study conducted in a VA outpatient treatment setting. The study is designed to test the feasibility of implementing a novel way of working with suicidal patients, the Collaborative Assessment and Management of Suicidality (CAMS). The primary purpose of the proposed project is to determine if it is possible to train clinicians working in the Mental Health Clinic at the Denver VA Medical Center (VAMC) to utilize this therapeutic framework. This project is extremely timely in relation to expectations of future increased clinical demands among potentially high-risk Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) veterans who may become suicidal in the years to come.

ELIGIBILITY:
Inclusion Criteria:

1. Suicidality endorsed during the regular Mental Health intake interview or at the time of admission.
2. Over the age of 18 years.
3. New or returning patients to the VA MHC.
4. Living within the larger Denver metropolitan region during the duration of the treatment.
5. Willing to travel to the ECHCS Denver VAMC at times other than scheduled therapy appointments to complete follow-up assessment measures.

Exclusion Criteria:

1. Psychosis that would interfere with an individual's ability to provide informed consent.
2. Imminent suicidality with the need for immediate psychiatric hospitalization, as defined above in the Background section, at the time of MH intake.
3. Current involuntary status for psychiatric hospitalization.
4. Inability to adequately respond to questions regarding the informed consent procedure. See Special Consent Issues section below.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Brenner, PhD, Principal Investigator — VISN 19 MIRECC
Locations (1):
- Visn 19 Mirecc, Denver, Colorado, United States